CLINICAL TRIAL: NCT04086329
Title: The Development of Minimally Invasive Nanosensor Technology to Quantify Mitochondrial Function in Human Muscle
Brief Title: Validation of Oxygen Nanosensor in Mitochondrial Myopathy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Zarazuela Zolkipli Cunningham, Principal Investigator, Children's Hospital of Philadelphia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-014130; 5U54NS078059-12 (NIH)
Record Dates: First submitted 2019-09-06; First posted 2019-09-11 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2024-12

CONDITIONS: Mitochondrial Myopathies; Mitochondrial Diseases
MeSH Terms: conditions — Mitochondrial Myopathies; Mitochondrial Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Affected MM Cases (Other): Key eligibility criteria for MM cases includes physically-capable adults (male and females, ages 18 to 65 years, inclusive) with genetically-confirmed MM with predominant symptoms of myopathy as expressed by exercise intolerance and muscle weakness and fatigue.
  Interventions: Device: Nanosensor
- Healthy Controls (Other): Adult healthy volunteers will be individually matched with corresponding MM cases based on age, biological sex, and body mass index.
  Interventions: Device: Nanosensor

INTERVENTIONS:
Device: Nanosensor — The purpose of the study is to test a device called a "nanosensor", which measures oxygen levels (a proxy of mitochondrial function) in muscle. The nanosensor has not been tested in humans nor has it been approved by the FDA.
  The study nanosensor measures 1.8 mm width x 6 mm length x 0.3 mm depth. Placement of the sterilized nanosensor involves a small incision for manual placement of the nanosensor in muscle forearm tissue.

SUMMARY:
Past mitochondrial disease treatment studies have been unsuccessful in determining treatment efficacy, and a major factor has been the lack of validated biomarkers in mitochondrial myopathy (MM). There is currently a growing number of potential new treatments to be tested through MM clinical intervention trials, which has created a pressing need for quantitative biomarkers that reliably reflect MM disease severity, progression, and therapeutic response.

The purpose of the study is to measure the efficacy of an electrochemical oxygen nanosensor to measure in vivo mitochondrial function in human muscle tissue, and its ability to discriminate MM patients from healthy volunteers. The data and results from this nanosensor study may contribute to current and future research, including improved diagnostic and therapeutic approaches for patients with mitochondrial disease.

DETAILED DESCRIPTION:
This is an investigational device clinical trial. MM cases and healthy volunteers will undergo nanosensor muscle oxygen measurement in exercised (dominant) forearm muscle during handgrip exercise. The same measurements will be repeated between 7 and 30 days later in the same forearm and at the same time of day for each participant to assess reproducibility.

After placement of the nanosensor in the forearm under local anesthesia, the primary outcome measure is nanosensor-muscle oxygen levels. The secondary outcome measure is an assessment of pain.

ELIGIBILITY:
Inclusion Criteria for Healthy Controls

1. Males and females, between the ages of 18 and 65 years, inclusive
2. Provide informed consent for study participation; able to understand and complete the protocol
3. Able to ambulate independently
4. Able to perform bicycle ergometry

Inclusion Criteria for MM Cases

1. Males and females, between the ages of 18 and 65 years, inclusive
2. Provide informed consent for study participation; able to understand and complete the protocol
3. Genetically-confirmed MM as defined by a diagnosis of primary mitochondrial disease (PMD) with predominant symptoms of myopathy as expressed by exercise intolerance and muscle weakness and fatigue.
4. Previously enrolled (or will enroll) in Children's Hospital of Philadelphia (CHOP) Institutional Review Board (IRB) study #08-006177 (Falk, PI) or CHOP IRB #16-013364 (Zolkipli, PI)
5. Able to ambulate independently
6. Able to perform bicycle ergometry

Exclusion Criteria for All Participants

Subjects will be excluded if any of the following apply:

1. Unable to provide informed consent and complete all study procedures, including ergometry
2. Non-ambulatory or unable to ambulate independently
3. Pregnant
4. Within 1 month of a recent hospital admission due to acute illness
5. Have severe cardiac disease as defined by an ejection fraction of less than 35% and New York Heart Association Functional Classification Class III; or severe pulmonary disease as defined by the need for supplemental O2 therapy or daytime ventilatory support
6. Have a tracheostomy
7. Have a known bleeding disorder and/or family history (first-degree relative) with a known bleeding disorder
8. Daily intake of aspirin or any other anti-platelet therapy which cannot be temporarily discontinued for medical reasons
9. a) Have known or suspected congenital or acquired immune deficiency; b) concurrent use of immunosuppressive drugs, including corticosteroids; c) past history of recurrent (more than 6 times per year) severe (required hospitalization) skin or soft tissue infections; d) history of infection or delayed wound healing after surgery or biopsy; e) known history of neutropenia with absolute neutrophil count less than 500/mm3
10. Undergo chronic steroid treatment as defined by daily oral intake (for more than 1 month) or have existing untreated endocrinopathies, such as hypothyroidism that caused acquired myopathy
11. Prone to hypertrophic scars and keloids
12. Have any other known inherited myopathy, such as Duchenne muscular dystrophy or congenital myopathy
13. Known allergy to lidocaine
14. Have a cognitive impairment that may prevent the ability to complete study procedures
15. Unable to comply with the requirements of the study protocol and/or unsuitable for the study for any reason, in the opinion of the principal investigator
16. Individuals from vulnerable populations (e.g., prisoners/detainees)
17. Participants who are unable to speak and/or read English (as participants will be required to be proficient to complete study procedures)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Nanosensor-muscle oxygen (Torr) levels | 60 minutes for data collection at each 2 study visits, up to 6 months.
  Nanosensor measured muscle O2 levels at baseline, during handgrip exercise and after exercise

SECONDARY OUTCOMES:
Pain and tolerability | At each 2 study visits, up to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Zarazuela Zolkipli-Cunningham, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No